CLINICAL TRIAL: NCT02186418
Title: Gene Transfer For Patients With Sickle Cell Disease Using A Gamma Globin Lentivirus Vector: An Open-Label Phase 1 / 2 Pilot Study
Brief Title: Gene Transfer for Patients With Sickle Cell Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision due to funding
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ARU-1801_Ph1_01
Record Dates: First submitted 2014-06-30; First posted 2014-07-10 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2023-07

CONDITIONS: Anemia, Sickle Cell
Keywords: sickle cell disease; sickle cell anemia; hemoglobinopathies; hematopoietic stem cell; gene transfer; gene therapy
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobinopathies

STUDY DESIGN:
Intervention Model Description: Gamma Globin Lentivirus Vector
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARU-1801 (Experimental): Autologous CD34+ hematopoietic stem cells transduced ex-vivo with gamma-globin lentiviral vector. Administered via IV infusion.
  Interventions: Genetic: ARU-1801

INTERVENTIONS:
Genetic: ARU-1801 — Autologous CD34+ hematopoietic stem cells transduced ex-vivo with a gamma-globin lentiviral vector
  * Subjects with sickle cell anemia will undergo hematopoietic stem cell procurement by bone marrow harvest or apheresis after mobilization with plerixafor
  * Reduced intensity chemotherapy conditioning with single dose melphalan will be used to facilitate engraftment of ex-vivo transduced cells.

SUMMARY:
The purpose of this Phase 1/2 study is to determine the feasibility and safety of stem cell collection and gamma-globin gene transfer, and success of gene correction in subjects with sickle cell disease

DETAILED DESCRIPTION:
This study will assess the feasibility, safety and efficacy of gene transfer using ARU-1801 (CD34+ cells transduced with the gamma-globin lentiviral vector). Gene transfer will occur ex-vivo into CD34+ enriched human bone marrow or plerixafor-mobilized peripheral blood hematopoietic stem cells (HSC) collected from subjects with severe sickle cell disease (SCD). Subjects will undergo reduced intensity chemotherapy conditioning with single-dose melphalan to facilitate engraftment of ex-vivo ARU-1801 via IV infusion. Subjects will return to the study site at regular intervals for follow-up for 2 years after the ARU-1801 infusion. It is anticipated that a separate long-term follow-up (LTFU) clinical study will be initiated, in which all subjects completing the 2 year study visit will be asked to consent and enroll, and will followed for a further 13 years.

ELIGIBILITY:
Inclusion Criteria

* Signed informed consent form.
* Has confirmed diagnosis of sickle cell disease (SCD)
* Has severe sickle cell disease, defined as one or more of the following:

  1. Minimum of two episodes of clinically diagnosed acute chest syndrome (ACS) requiring hospital admission, or one life threatening episode of ACS requiring intensive care unit (ICU) admission for exchange transfusion and/or intubation, or frequent ACS episodes which necessitate treatment with chronic transfusion therapy.
  2. Frequent painful vaso-occlusive episodes (VOEs) which significantly interfere with normal life activities, defined as a history of 2 or more severe acute sickle pain events per year requiring additional treatment at a medical facility outside of home pain management over the preceding 2-year period prior to study enrollment, or that necessitate chronic transfusion therapy.
  3. Subjects on chronic transfusion therapy for severe disease symptoms other than those listed above, and which interfere with normal life activities.
* Has failed hydroxyurea therapy, was unable to tolerate hydroxyurea therapy, or has actively made the choice to not take the recommended daily hydroxyurea advised for severe disease (Note: must be off hydroxyurea therapy for 2 months prior to stem cell collection). If refusing hydroxyurea, the subject must document that they have been educated about the benefits and continue to refuse the treatment. Patients placed on chronic transfusion therapy instead of hydroxyurea for severe disease are eligible. Subjects unable to take hydroxyurea due to financial or safety monitoring constraints are eligible.
* Has adequate functional status and organ function as determined at Screening.

Exclusion Criteria

* Female subjects who are pregnant or lactating/breastfeeding.
* Female subjects who are not surgically sterile, postmenopausal or who refuse to practice effective method of birth control as determined by the Investigator for one year after receiving the study drug. Women must also agree not to breastfeed for 1 year after receiving the study drug.
* Any participant of reproductive potential who refuses to agree to use an appropriate contraceptive method determined by the Investigator, for 1 year after receiving the study drug.
* Patients with an active malignant disease or receiving treatment for any type of cancer (except squamous cell carcinoma, basal cell carcinoma, or carcinoma in situ of the skin).
* Current diagnosis or history of hepatitis B, hepatitis C, or HIV.
* Has received another study drug within 30 days, or 5 half-lives of the last dose (whichever is longer), prior to screening.
* Has severe obstruction, restriction or diffusion defect on pulmonary function tests.
* Has uncontrolled bacterial, viral or fungal infections within 1 month prior to starting the conditioning part of the study. Subjects with fever should wait for symptoms to resolve before starting the conditioning part of the study.
* Has a history of stroke or is at moderate to high risk of primary stroke (eg receiving chronic transfusions or hydroxyurea for primary prevention of stroke; has severe cerebral vasculopathy defined as moderate stenosis in >2 arterial segments; and/or has sever stenosis/occlusion in ≤2 segments in the polygon of Willis or presence of Moyamoya-like disease).
* Patients with alpha thalassemia sickle cell disease.
* Has previous liver biopsy showing cirrhosis, bridging hepatic fibrosis, or active hepatitis; or has received chronic transfusions and has previous evidence of iron overload and evidence of liver fibrosis by noninvasive liver imaging.
* Has a matched sibling donor, unless the subject has declined this option or this option is not feasible. Documentation must be included as part of the informed consent process for subjects who decline this option.
* Has a known hypersensitivity to any study treatments (e.g. melphalan, plerixafor).

Other protocol-defined inclusion-exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Grade 3 allergic reaction | From infusion (Day 0) to 15 years
  Incidence of Grade 3 allergic reaction associated with infusion of transduced cell product
Incidence of Grade 4 infection | From infusion (Day 0) to 15 years
  Incidence of Grade 4 infection following infusion of transduced cell product uncontrolled for ≥14 days
Incidence of Grade 4 neutropenia | From date of chemotherapy clearance visit to 15 years post-infusion of transduced cells
  Incidence of Grade 4 neutropenia lasting >1 month following melphalan
Incidence of Grade 3 or 4 organ toxicity | From screening to 15 years post-infusion of transduced cells
  Incidence of Grade 3 or 4 organ toxicity attributable to study procedures
Incidence of Adverse Events (AEs) | From screening to 15 years post-infusion of transduced cells
Incidence of Serious Adverse Events (SAEs) | From screening to 15 years post-infusion of transduced cells
Incidence of death due to study procedures | From screening to 15 years post-infusion of transduced cells
Incidence of hematological malignancy | From infusion (Day 0) to 15 years
  Incidence of hematological malignancy due to vector insertion
Incidence of hematological cancer | From screening to 15 years post-infusion of transduced cells
  Incidence of hematological cancer related to investigational product or study medications/procedures
Time to neutrophil recovery | From ≥36 hours before Day 0 to 2 years post-infusion of transduced cells
  Number of days from melphalan-induced nadir to the first of 3 consecutive absolute neutrophil counts ≥500 cells/µL
Time to platelet recovery | From ≥36 hours before Day 0 to 2 years post-infusion of transduced cells
  Number of days from melphalan-induced nadir to the first of 3 consecutive platelet counts >50,000 cells/µL and independent of platelet transfusion for ≥7 days consecutive days.
≥8x10⁶kg viable CD34+ cells | Up to Year 2
  Number of subjects with a total number of CD34+ cells recovered from all collections combined (mobilized peripheral blood and bone marrow) of at least ≥8x10⁶kg viable CD34+ cells
≥4x10⁶ CD34+ cells/kg body weight transduced | Up to Year 2
  Proportion of subjects for which a minimum of 4x10⁵ CD34+ cells/kg body weight from all collections combined have been successfully transduced
Bone marrow aspirates with ≥1% gene-marked cells | Infusion (Day 0) to 1 year
  Number of subjects with bone marrow aspirates at 1-year post-infusion with ≥1% gene-marked cells

SECONDARY OUTCOMES:
Quantity of Hb (hemoglobin) subtypes | Months 6, 12, 18, 24 and year 3, 4, 5
  Quantification of HbF^G16D and other Hb subtypes, including HbF (endogenous), HbS, adult Hb (HbA), HbA2 and, if applicable, HbC and HbE
Change in proportion of antisickling/sickling hemoglobin | Baseline to Month 6 through 12
  Change in the proportion of antisickling/sickling hemoglobin ([HbF+HbF^G16D+HbA2]/HbS) in months 6-12 post-transplantation compared to baseline
Percentage of F-RBC (fetal hemoglobin content in red blood cells) | Months 6, 12, 18, 24, 36
  Measured by flow cytometry
Percentage of F-retics (fetal hemoglobin content in reticulocytes) | Months 6, 12, 18, 24, 36
  Measured by flow cytometry
Presence of vector copies in white blood cell fraction | Days 30, 60, 90, Months 4, 5, 6, 9, 12, 18, 21, 24
Presence of vector copies in bone marrow | Prior to ARU-1801 infusion, month 6, 12, 18, 24 and 36
  Measured by qPCR and DNA
Presence of gene-marked colony-forming unit cells (CFU-c) in bone marrow (BM) indicting gene transfer | Prior to ARU-1801 infusion, month 6, 12, 18, 24 and 36
  Measured by CFU-c assay by qPCR on individual CFU-c
Number of annualized vaso-occlusive episodes (VOEs) pre-transplant versus post-transplant | Baseline to year 15
  Change in disease severity
Frequency of opioid use pre-transplant versus post-transplant | Baseline to year 15
  Change in disease severity
Change in QoL (Quality of Life) | Baseline, month 4, 5, 6, 12 and 24 and year 3, 4, 5
  Measured by adult sickle cell quality of life measurement (ASCQ-Me®)

CONTACTS AND LOCATIONS:
Overall Officials: Stella M. Davies, MB BS, PhD, MRCP, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grimley M, Davies SM, Shrestha A, Shova A, Asnani M, Kent M, Sayani F, Quinn CT, Niss O, Lutzko C, Mehta PA, Khandelwal P, Little C, Chandra S, Felker S, Chi M, Kalfa TA, Knight-Madden J, Arumugam PI, Ramos KN, Witting S, Latham T, Bushman FD, Malik P. Lentiviral gene therapy with reduced-intensity conditioning for sickle cell disease: a phase 1/2 trial. Nat Med. 2025 Jul;31(7):2204-2212. doi: 10.1038/s41591-025-03662-2. Epub 2025 May 26. PMID 40419809

DOCUMENTS (1):
  • Study Protocol (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT02186418/Prot_000.pdf